CLINICAL TRIAL: NCT04069130
Title: An Open-Label Study to Assess the Absorption, Distribution, Metabolism and Excretion, Including the Mass Balance Recovery, Metabolite Profiling and Identification, of [14C] Labelled BIA 5-1058 Following a Single Oral Dose Administration in Healthy Male Subjects
Brief Title: Absorption, Distribution, Metabolism and Excretion of [14C] Labelled BIA 5-1058
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA-51058-119
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BIA 5 (Experimental): single oral dose of 400 mg as an oral capsule
  Interventions: Drug: 400 mg of BIA 5-1058

INTERVENTIONS:
Drug: 400 mg of BIA 5-1058 — 1 x 400 mg capsule Oral, Fasted

SUMMARY:
The purpose of the study is to determine the mass balance recovery in expired air, urine and faeces after a single oral dose of 400 mg 14C-labeled BIA 5-1058; to provide plasma, urine and faecal samples for metabolite profiling and structural identification; and determine the routes and rates of elimination of [14C]-BIA 5-1058

DETAILED DESCRIPTION:
This is a Phase 1, single-dose, single-centre, single period, open-label, absorption, distribution, metabolism and excretion study in 8 healthy adult male subjects. Subjects will receive a single oral dose of 400 mg [14C]-BIA 5-1058, containing not more than (NMT) 4.6 MBq (124 µCi) 14C, as an oral capsule. Subjects will be screened for eligibility to participate in the study between 28 and 2 days before dosing. Eligible subjects will be admitted to the clinical unit on the morning of Day -1 prior to investigational medicinal product (IMP) administration. Subjects will be dosed on the morning of Day 1 after an overnight fast of at least 10 hours and will remain resident in the clinic until up to 336 h after dosing (up to Day 15). Blood, urine, faeces and expired air will be collected at predefined time points for mass balance and PK analysis. It is planned that subjects will be released as a group when all subjects have achieved a mass balance cumulative recovery of >90% or if <1% of the dose administered has been collected in urine, faeces and expired air within 2 separate, consecutive 24 h periods. This may result in the subjects being discharged as a group prior to completion of the planned residency period. Once the discharge criteria or the planned residency period has been achieved, collection of all samples (blood, urine, faeces, and expired air) will be stopped and the subjects will undergo discharge assessments. Subjects who have not met the mass balance discharge criteria on Day 15 will return to the clinical unit for up to five further 24-hour residency periods (Days 21-22 [±1 day], 28-29 [±1 day], 42-43 [±2 days], 56-57 [±2 days] and 77-78 [±3 days]) to collect blood samples for PK analysis and urine and faeces samples for analysis of total radioactivity. If the parent and metabolite are below the limit of quantification at any of these visits, subsequent return visits may be cancelled. If by Day 78, levels are not below the limit of quantification or if the additional 24 h residency periods are not considered appropriate or necessary, then home collections of urine and/or faeces may be requested at the discretion of the investigator for individual subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males;
* Age 30 to 65 years of age, inclusive;
* Body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive;
* Normal resting supine BP (Systolic BP: 90-140 mmHg [age 18-45] 90 160 mmHg [age >45], Diastolic BP: 40-90 mmHg) and heart rate: 40-90 bpm (age 18-45) 50-90 bpm (age >45) or showing no clinically relevant deviation as judged by the investigator or delegate;
* Digital (12-lead) ECG recording without signs of clinically relevant pathology or showing no clinically relevant deviations as judged by the investigator or delegate;
* All values for clinical laboratory tests of blood and urine within the normal range or showing no clinically relevant deviations as judged by the investigator or delegate;
* Must be willing and able to communicate and participate in the whole study;
* Must have regular bowel movements (ie, average stool production of between ≥1 every 2 days and ≤3 stools per day);
* Must provide written informed consent;
* Must agree to adhere to the contraception requirements

Exclusion Criteria:

* Females;
* Subjects who have received any IMP in a clinical research study within the previous 90 days prior to Day 1 of the study;
* Subjects who are study site employees, or immediate family members of a study site or sponsor employee;
* Subjects who have previously received BIA 5-1058 (including participation in QCL118167);
* History of any drug or alcohol abuse in the past 2 years;
* Regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type);
* Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening and admission;
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months;
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study;
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening;
* Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator (laboratory parameters are listed in Appendix 2);
* Positive drugs of abuse test result;
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results;
* An estimated creatinine clearance of <90 mL/min based on creatinine clearance calculation using the Cockcroft-Gault equation and normalised to an average surface area of 1.73 m2;
* Clinically significant history of cardiovascular, renal, hepatic, respiratory and particularly GI disease, especially peptic ulceration, GI bleeding, ulcerative colitis, Crohn's Disease or Irritable Bowel Syndrome, as judged by the investigator or sub investigator;
* Frequent headaches and/or migraine, recurrent nausea, and/or vomiting (more than twice a month);
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients;
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active;
* Donation or loss of greater than 400 mL of blood within the previous 3 months;
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than 2 g paracetamol per day) or herbal remedies in the 14 days before IMP administration. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor;
* Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Ae(urine) - amount excreted in urine | Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Calculation of Mass balance of total radioactivity
Ae(faeces) - amount excreted in faeces | Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Calculation of Mass balance of total radioactivity
Ae(expired air) - amount excreted in expired air | Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Calculation of Mass balance of total radioactivity
Ae(total) - amount excreted in urine, faeces and expired air combined | Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Calculation of Mass balance of total radioactivity
CumAe(urine) - cumulative amount excreted in urine | Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Calculation of Mass balance of total radioactivity
CumAe(faeces) - cumulative amount excreted in faeces | Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Calculation of Mass balance of total radioactivity
CumAe(expired air) - cumulative amount excreted in expired air | Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Calculation of Mass balance of total radioactivity
CumAe(total) - cumulative amount excreted in urine, faeces and expired air combined | Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Calculation of Mass balance of total radioactivity
%Ae(urine) - amount excreted in urine expressed as a percentage of the administered dose | Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Calculation of Mass balance of total radioactivity
%Ae(faeces) - amount excreted in faeces expressed as a percentage of the administered dose | Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Calculation of Mass balance of total radioactivity
%Ae(expired air) - amount excreted in expired air expressed as a percentage of the administered dose | Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Calculation of Mass balance of total radioactivity
%Ae(total) - amount excreted in urine, faeces and expired air combined expressed as a percentage of the administered dose | Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Calculation of Mass balance of total radioactivity
Cum%Ae(urine) - cumulative amount excreted in urine expressed as a percentage of the administered dose | Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Calculation of Mass balance of total radioactivity
Cum%Ae(faeces) - cumulative amount excreted in faeces expressed as a percentage of the administered dose | Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Calculation of Mass balance of total radioactivity
Cum %Ae(expired air) - cumulative amount excreted in expired air expressed as a percentage of the administered dose | Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Calculation of Mass balance of total radioactivity
Cum %Ae(total) - cumulative amount excreted in urine, faeces and expired air combined expressed as a percentage of the administered dose | Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Calculation of Mass balance of total radioactivity
Tmax- the time from dosing at which Cmax was apparent | Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Pharmacokinetic Data Analysis
Cmax - maximum observed concentration | Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Pharmacokinetic Data Analysis
C24 - plasma concentration at 24 h | Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Pharmacokinetic Data Analysis
AUC(0-last) - area under the curve from 0 time to last measurable concentration | Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Pharmacokinetic Data Analysis
AUC(0-inf) - area under the curve from 0 time extrapolated to infinity | Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Pharmacokinetic Data Analysis
AUC%extrap - percentage of AUC(0-inf) extrapolated beyond last measured time point | Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Pharmacokinetic Data Analysis
Lambda-z - the slope of the apparent elimination phase | Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Pharmacokinetic Data Analysis
Kel - elimination rate constant | Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Pharmacokinetic Data Analysis
T1/2 - the apparent elimination half-life | Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Pharmacokinetic Data Analysis
CL/F - total body clearance after extravascular administration (for BIA 5 1058 in plasma only) | Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Pharmacokinetic Data Analysis
Vz/F - apparent volume of distribution based on the terminal phase after extravascular administration (for BIA 5 1058 in plasma only). | Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15.
  Pharmacokinetic Data Analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No